CLINICAL TRIAL: NCT01504724
Title: Effect of Adjunctive Intravitreal Bevacizumab Before Panretinal Photocoagulation in Macular Thickness and Retinal Nerve Fiber Layer Thickness
Brief Title: Effect of the Adjunctive IVB Before PRP
Acronym: IVB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Park, Clinical professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVB and PRP
Record Dates: First submitted 2012-01-01; First posted 2012-01-05 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Retinopathy
Keywords: central macular thickness
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVB group (Experimental): Patients were treated with IVB injections approximately within 1 week before the first PRP. Then patients had PRP, which was done in three sessions at weeks 0, 1, and 2 according to ETDRS guidelines. The superior, inferior, and nasal and temporal areas were treated sequentially.
  Interventions: Drug: bevacizumab
- only PRP group (No Intervention): Patients had PRP, which was done in three sessions at weeks 0, 1, and 2 according to ETDRS guidelines. The superior, inferior, and nasal and temporal areas were treated sequentially.

INTERVENTIONS:
Drug: bevacizumab — intravitreal bevacizumab injection (1.25 mg/0.05 mL) was done 4.0 mm posterior to the corneal limbus using a 30-gauge needle after topical anesthesia
  Other Names: Avastin; Genentech, Inc., South San Francisco, CA, USA
  Arms: IVB group

SUMMARY:
This study is to investigate the effect of adjunctive intravitreal bevacizumab (IVB) before panretinal photocoagulation (PRP) compared with only PRP on central macular thickness and retinal nerve fiber layer thickness in patients with severe diabetic retinopathy without macular edema.

DETAILED DESCRIPTION:
This prospective randomized study included 30 patients (60 eyes) with severe nonproliferative diabetic retinopathy or non-high-risk proliferative diabetic retinopathy. They had weekly PRP treatments in 3 sessions and they were randomly assigned to IVB group who had adjunctive IVB within 1 week before first PRP and control group who had only PRP. CMT, RNFL, and best-corrected visual acuity (BCVA) were measured

ELIGIBILITY:
Inclusion Criteria:

* patients with severe NPDR or early PDR without macular edema
* best-corrected visual acuity (BCVA) of 20/25 or better
* patients who were followed up for at least 6 months after the first PRP.

Exclusion Criteria:

* patients with retinal or choroidal diseases except diabetic retinopathy
* contraindications to fluorescein angiography (FA) or bevacizumab
* patients who had previous treatments including anti-angiogenic medications and laser photocoagulation
* patients with previous vitrectomy
* patients with uncontrolled hypertension, a recent myocardial infarction or cerebral vascular accidents.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Central macular thickness | 6 months after first PRP session
  central macular thickness measured by Cirrus HD optical coherence tomography

SECONDARY OUTCOMES:
Retinal nerve fiber layer thickness | 6 months after first PRP session
  retinal nerve fiber layer thickness measured by Cirrus HD optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ho Park, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Dong Ho Park, Daegu, South Korea

REFERENCES:
- [Background] Jo YJ, Heo DW, Shin YI, Kim JY. Diurnal variation of retina thickness measured with time domain and spectral domain optical coherence tomography in healthy subjects. Invest Ophthalmol Vis Sci. 2011 Aug 17;52(9):6497-500. doi: 10.1167/iovs.11-7403. PMID 21705686